CLINICAL TRIAL: NCT01064141
Title: Immunogenicity and Safety of CYD Dengue Vaccine in Healthy Toddlers Aged 12 to 15 Months in the Philippines
Brief Title: A Study of Dengue Vaccine in Healthy Toddlers Aged 12 to 15 Months in the Philippines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD08; UTN: U1111-1111-5855 (Other: WHO)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; CYD Dengue Vaccine; Toddlers
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Dengue Vaccine Group (Experimental): Participants will receive CYD Dengue vaccine as Visits 1 and 2.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus
- Group 2: Control Group (Active Comparator): Participants will receive Control Vaccines. (Varicella at Visit 1 and Hepatitis A at Visit 2)
  Interventions: Biological: OKAVAX®:Attenuated live varicella-zoster virus and AVAXIM® 80U: Hepatitis A virus Vaccines
- Group 3: Co-administration Group (Experimental): Participants will receive CYD Dengue vaccine and childhood vaccines at Visit 1 and CYD Dengue vaccine at Visit 2.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus and Childhood vaccines
- Group 4: Sequential Administration Group (Experimental): Participants will receive CYD Dengue vaccine and a Placebo vaccine at Visit 1 and CYD Dengue vaccine at Visit 2.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus and NaCl (Placebo)

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: Group 1: Dengue Vaccine Group
Biological: OKAVAX®:Attenuated live varicella-zoster virus and AVAXIM® 80U: Hepatitis A virus Vaccines — 0.5 mL, Subcutaneous and 0.5 mL, Intravascular
  Other Names: OKAVAX®; AVAXIM® 80U
  Arms: Group 2: Control Group
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus and Childhood vaccines — 0.5 mL, Subcutaneous and 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine; TRIMOVAX®
  Arms: Group 3: Co-administration Group
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3 and 4 virus and NaCl (Placebo) — 0.5 mL Subcutaneous and 0.5 mL Subcutaneous
  Other Names: CYD Dengue Vaccine; NaCl 0.9% (Placebo)
  Arms: Group 4: Sequential Administration Group

SUMMARY:
The purpose of this study is to investigate the potential for co-administration of the first dose of CYD Dengue vaccine with childhood vaccination.

Primary Objectives:

* To describe the safety of CYD Dengue vaccine after each dose; first dose given alone or coadministered with childhood vaccines.

Secondary Objectives:

* To describe the immunogenicity of CYD Dengue vaccine after each dose; first dose given alone or co-administered with childhood vaccines.

DETAILED DESCRIPTION:
Participants will be enrolled in a 3-step enrollment and randomized to 1 of 4 treatment groups. Groups 1 and 2 will receive 5 vaccinations, and Groups 3 and 4 will received 6 vaccinations (childhood vaccines or placebo co-administered with the first dose of CYD Dengue vaccine in 2 separate arms). All toddlers will receive a pentavalent acellular pertussis combination vaccine or Combo (PENTAXIM®), planned approximately 10 months after enrollment.

ELIGIBILITY:
Inclusion Criteria :

* Toddler in good health based on medical history and medical examination
* Toddler aged 12 to 15 months on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Provision of informed consent form signed by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations)
* Participant and parent/delegate able to attend all scheduled visits and comply with all trial procedures
* Completion of previous vaccination program according to the national immunization schedule, except for measles

Exclusion Criteria :

* Family members from the Investigator or from the staff involved in the trial
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of central nervous system disorder or disease, including seizures
* History of varicella, measles, mumps, rubella and hepatitis A; confirmed either clinically, serologically, or microbiologically
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion
* Previous vaccination against measles-mumps-rubella, hepatitis A or varicella
* Previous vaccination against flavivirus diseases
* Known systemic hypersensitivity to any of the components of the vaccines, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Planned participation in another clinical trial during the present trial period
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination
* Human immunodeficiency virus (HIV) seropositivity in the blood sample taken at screening
* Clinically significant laboratory abnormalities, as judged by the Investigator, in blood sample taken at screening

Temporary exclusions: vaccination postponed until the condition is resolved:

* Febrile illness (temperature ≥ 38°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Receipt of oral or injected antibiotic therapy within 72 hours prior to the vaccination visit
* Any vaccination received in the 4 weeks preceding vaccination

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety in terms of solicited and unsolicited adverse events after primary administration of CYD Dengue vaccine. | 28 days after each Dengue vaccination and entire study duration

SECONDARY OUTCOMES:
To provide information concerning the immunogenicity of CYD Dengue vaccine after each dose of primary vaccination. | Day 28 after each Dengue vaccination
To provide information concerning the immunogenicity of childhood vaccines after primary vaccination. | Day 28 after post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- San Pablo, Philippines

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com